CLINICAL TRIAL: NCT00817466
Title: Bronchiolitis All-study, SE-Norway What is the Optimal Inhalation Treatment for Children 0-12 Months With Acute Bronchiolitis?
Brief Title: Bronchiolitis All-study, SE-Norway
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Ostfold University College (Other); Vestre Viken Hospital Trust (Other); Sykehuset i Vestfold HF (Other); Sykehuset Telemark (Other Government); Sorlandet Hospital HF (Other Government); Sykehuset Innlandet HF (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT 2009-012667-34
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; infants; racemic adrenaline; inhalations; treatment
MeSH Terms: conditions — Bronchiolitis; Respiratory Aspiration | interventions — Racepinephrine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Racemic adrenaline, fixed intervals (Experimental): Active drug with fixed intervals of inhalation, adjusted at least every 24h.
  Interventions: Drug: Racemic adrenaline
- Racemic adrenalin, on demand (Experimental): Racemic adrenaline, inhalations on demand (max every 2 hrs)
  Interventions: Drug: Racemic adrenaline
- Saline, fixed intervals (Active Comparator): Saline inhalation fixed intervals, adjusted at least every 24 hrs
  Interventions: Drug: Isotonic saline
- saline on demand (Active Comparator): Saline inhalations on demand, max every 2 hrs, adjusted every 12 hrs
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Racemic adrenaline — For inhalation.
  Dosing (as in previous study):
  1) 0,1ml<5kg, 0,15ml 5-6,9kg, 0,20ml 7-9,9kg, 0,25ml >10kg of racemic adrenaline 20mg/ml diluted in 2ml NaCl 9mg/ml.3
  Maximum 12 inhalations/24 hours. One bottle (10ml) per patient. The bottles will be marked with the name of the study and a randomisation number.
  Other Names: Racemic adrenaline, racemic epinephrine, S2, vaponefrin, micronefrin
  Arms: Racemic adrenalin, on demand; Racemic adrenaline, fixed intervals
Drug: Isotonic saline — 2ml NaCl 9mg/ml.
  Other Names: Isotonic saline. NaCl 0,9%. NaCl 9mg/ml.
  Arms: Saline, fixed intervals; saline on demand

SUMMARY:
Bronchiolitis is a common lower respiratory disease typically affecting infants and children generally younger than 2 years of age. The disease leads to hospital admissions, is a major cause for hospitalisation of young children and infants during winter epidemics, may be severe sometimes requiring ventilatory support and rarely death. The clinical disease as described by Court is characterised by nasal flaring, tachypnoea, dyspnoea, chest recessions, crepitations and sometimes sibiliations. Respiratory Syncytial virus is the most common cause, but also other respiratory vira may cause the disease. Bronchiolitis is a well known risk factor of asthma development in childhood1,2.

Management is generally supportive, whereas symptom reducing therapy is debated with no international consensus. Furthermore, there are many unresolved questions related to the prognosis of bronchiolitis, its role in development of chronic lung disease in particular regarding the association between early bronchiolitis and asthma development. The present project will particularly focus on: 1)Treatment efficacy related to various outcomes during active disease, 2) retrospectively assess treatment efficacy in relation to later development of allergic disease, 3) assess the role between different vira and asthma prognosis as well as 4) identify possible prognostic factors involved in the progression from bronchiolitis to further airways disease.

DETAILED DESCRIPTION:
OVERALL AIMS OF THE STUDY:

1. To compare the efficacy of two common treatments by determining whether inhalation treatment with racemic adrenaline is more effective than saline inhalations in acute bronchiolitis in children younger than 12 months throughout an hospital admission, as well as to define the optimal inhalation treatment intervals.
2. To identify clinical and virological risk factors for development of persisting obstructive airways disease after an initial bronchiolitis, and to assess if specific vira or subsequent asthma development influences the efficacy of bronchiolitis management.
3. To assess whether hospital admissions for bronchiolitis has increased in parallel with the increase in childhood asthma seen in the last 10-15 years.

METHODS AND STUDY PROGRESSION

Design:

This multicenter study will be performed after initial appropriate common training by all participating.

1. Treatment study: The study will follow the standard operating procedure of Good Clinical Practice, including a clinical monitor from Oslo University Hospital, Ullevål who will provide study quality assurance in all centers. Two main groups randomised into RA vs saline, each divided into two arms of the active drug/NaCl groups: fixed or on demand inhalations. The trial will be double blinded by the pharmacy. One glass with sufficient medication for the entire hospital stay will be designated per patient throughout. No cross-over. Outcomes will be analysed by intention to treat, with treatment given and recorded throughout the hospital admission. No interim analyses are planned since the study compares two established treatment modalities used for the last decades.

   Inclusion into the treatment study provides the basis for the follow-up (prognosis) part of the study.
2. Prognosis: 18 months follow-up study (clinical assessment) of all subjects in the treatment study.The prognosis study will also retrospectively answer whether treatment efficacy depend upon later allergic disease development.
3. Epidemiology: a retrospective chart study for hospital admissions for bronchiolitis within populations referred to the collaborating centres in HSØ from 1995-2009

Methods:

a. Treatment: Randomisation: block randomisation. Randomization will be performed by computer programs by the ORAACLE statistician, and provided to the Pharmacy preparing and labeling the vials for each patient.

Treatment: Nebulised racemic adrenaline vs saline throughout the hospital stay. Inhalations given on demand (parents/nurse) vs fixed x 4--12. Open saline inhalations may be given at any time, other inhalations is not allowed. Neither is systemic corticosteroids (which is not a proper treatment for acute bronchiolitis, according to Norwegian guidelines). All other treatment will be given according to usual local practice.

Study end-points:

1. Treatment study: Completion of the study at discharge + possible re-admission according to protocol. Need for intensive care management or assisted ventilation (continuous CPAP-Ventilator) in which conventional management will be given. Treatment failure when the child is assessed severely ill and in need of open label treatment. These data will be recorded and analysed to see if there is a difference between the two treatment groups. We expect a small number of drop-outs, which should not make it necessary to expand the study above our goal of 500 patients.
2. Prognosis study: Number of children with recurrent bronchial obstruction (wheeze), secondary: asthma diagnosis, the "Oslo severity score".
3. Hospital admissions first time, secondary: re-admissions or multiple admissions

Methods:

Clinical scores will be assessed before and 30 minutes after inhalation the first time, and subsequently once a day during ordinary doctor visit.

Global clinical assessment completed by nurses and parents will be done every morning and evening until discharge. Time at start, end and hours with naso-gastric tube feeding as well need for supplementary oxygen will be recorded daily and complications and adverse event will be recorded as they appear.

Nasopharynx aspiration is done at inclusion and is analysed by local routine, usually within 24 hours (except Sundays). Half of the aspirate will be frozen for batch PCR analyses at the virological laboratory (Oslo University Hospital) after all patients are enrolled.

Blood tests are sampled at inclusion. General analyses (see table 6) and sample to biobank for epigenetic analyses.

Saliva are sampled at inclusion and the following morning. Deemed fit for discharge will be decided by the attending physician. Minimum requirement is clinical score 3 or less at least 2 hours after last inhalation.

Urine tests are sampled at inclusion. Will be analysed at leukotrienes and arachidonic acid metabolites (eoxines) and other relevant inflammatory and infection markers.

Outcomes measured upon inclusion, after first inhalation (clinical score) as well as throughout the hospital stay according to flow-chart.

Main outcome: No of hours before deemed fit for discharge from hospital

Secondary:

Need for feeding support (no. of hours) Need for supplementary oxygen. Clinical score throughout admission Complications (presence of and time to confirmed) such as atelectasis Global assessments (parents and nurses) Need for ICU treatment Data from each hospital will in addition to collated data analysis be assessed independently.

Illness caused by different vira will be compared in regard to treatment efficacy.

b. Prognosis: This follow-up-study will be performed in collaboration between the principal investigator and the collaborating physicians at the local paediatric departments. The clinical follow-up visit includes a structured parental interview, application of the "Oslo severity score"20 for obstructive airways disease, assessment of atopic eczema and rhinitis, skin prick test as well as blood sampling for analyses including IgE and DNA for epigenetic studies (see table 4) .

c. Epidemiology: Retrospective study of all children 0-18 months admitted to hospital with the diagnosis of bronchiolitis. The study will mainly be a hospital registry study, but with 20% random chart scrutiny to ensure appropriateness of diagnosis.

Ammendment: Two further substudies were included;

a) Quality of life after bronchiolitis b) A population-based control group of 241 children from Oslo and Fredrikstad were included.

1. Description Quality of Life:

   ITQOL was sent to all children included in the RCT cohort, as well as the control group (see below) 6-9 months after enrollement in the study, as well as prior to the 18-month follow-up study.

   Main objective: To assess if quality of life after acute bronchiolitis in infancy is associated with development of persisting obstructive airways disease or allergic disease in early childhood.

   Specific aim 1: What is the quality of life in infants and parents 6 and 18 months after hospital admission for acute bronchiolitis? Specific aim 2: Is quality of life in infants and their parents 6 and 18 months after hospital admission for acute bronchiolitis related to recurrent or persisting obstructive airways symptoms? Specific aim 3: Is a possible association between quality of life and persistent obstructive airways disease modified by allergic sensitisation, gender or type of virus infection during the bronciolitis
2. Description Control group:

Since we established the "Bronchiolitis" cohort of children admitted to hospital for acute bronchiolitis, the prognostic perspective of this three-phase study has gained increasing focus. This relates in particular to immunological influence of different viral agents during the acute disease, as well as Quality of Life and the role of early "stress" in relation to development of allergic diseases in children with as well as without acute bronchiolitis in early life.

The aims are to assess physiological, immunological, environmental and "stress" (including psychosocial) factors in the development of allergic diseases, including asthma, atopic eczema, allergic rhinitis and allergies in children who have been hospital admitted due to acute bronchiolitis in infancy as well as children of the same age who have not been admitted for bronchiolitis.

Control children will be consecutively included at 2 Well-baby clinics in Fredrikstad and Oslo, respectively, total number 150 (100 + 150, respectively) ensuring similar variability of demographic data (age and ethnic background) as the enrolled bronchiolitis children. Inclusion will be assessed mid-way for adequate demographic variability.

Inclusion criteria: children 1- 11 months (inclusive) of age presenting to the Well-Baby Clinics, Exclusion criteria: Significant cardiac, previous severe respiratory disease, neurologic, immunologic, oncologic or other disease that may significantly influence the outcomes, including Down's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* children 0 inclusive 11 months admitted to the hospital with symptoms and signs of acute bronchiolitis during the winter season of 2009-11.
* bronchiolitis as defined on clinical criteria by SDM Court (Post graduate medical journal 1973).
* Clinical score of 4 or more (Kristjansson, Arch.Dis.Child. 1993)

Exclusion criteria:

* Use of regular inhaled corticosteroids.
* Use of systemic or inhaled corticosteroids within the last 4 weeks.
* Significant cardiac, previous severe or persisting (>4 weeks) respiratory disease, neurologic, immunologic, oncologic or other disease that may significantly influence the outcomes, including Down's syndrome. Prematurity per se is not a reason for exclusion.
* One single previous mild-moderate episode suspect of bronchial obstruction is not an exclusion criterion, >1 are.

Max Age: 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
No of hours before deemed fit for discharge from hospital | Throughout the hospital stay

SECONDARY OUTCOMES:
Clinical status (by parents as well as nurses) every 12 hrs | prior to inhalation every morning and evening
Need for feeding support (no. of hours) | Throughout the hospital stay.
Need for supplementary oxygen. | Throughout the hospital stay.
Clinical score measured by doctor | Throughout the hospital stay. Daily before and 30min after inhalation in daytime.

CONTACTS AND LOCATIONS:
Overall Officials: Karin C. Lødrup Carlsen, MD,pHD, Study Director — Ullevål University Hospital HF; Håvard O Skjerven, MD, Principal Investigator — Ullevål University Hospital HF
Locations (9):
- Norway (9):
  - Sykehuset Buskerud, Vestre Viken, Drammen, Buskerud
  - Sykehuset Innlandet, Elverum, Elverum, Hedmark
  - Sykehuset Innlandet, Lillehammer, Lillehammer, Oppland
  - Oslo University Hospital, Rikshospitalet, Oslo, Oslo County
  - Sykehuset Telemark, Skien, Skien, Telemark
  - Sørlandet sykehus HF, Kristiansand, Kristiansand, Vest-Agder
  - Sykehuset Vestfold, Tønsberg, Tønsberg, Vestfold
  - Ullevaal University Hospital, department of Paediatrics, Oslo
  - Sykehuset Østfold, Fredrikstad, Fredrikstad, Østfold fylke

REFERENCES:
- [Derived] Skjerven HO, Hunderi JOG, Carlsen KH, Rolfsjord LB, Nordhagen L, Berents TL, Bains KES, Buchmann M, Carlsen KCL. Allergic sensitisation in infants younger than one year of age. Pediatr Allergy Immunol. 2020 Feb;31(2):203-206. doi: 10.1111/pai.13135. Epub 2019 Nov 7. No abstract available. PMID 31594030
- [Derived] Gjengsto Hunderi JO, Lodrup Carlsen KC, Rolfsjord LB, Carlsen KH, Mowinckel P, Skjerven HO. Parental severity assessment predicts supportive care in infant bronchiolitis. Acta Paediatr. 2019 Jan;108(1):131-137. doi: 10.1111/apa.14443. Epub 2018 Jun 29. PMID 29889987
- [Derived] Berents TL, Carlsen KCL, Mowinckel P, Skjerven HO, Rolfsjord LB, Nordhagen LS, Kvenshagen B, Hunderi JOG, Bradley M, Thorsby PM, Carlsen KH, Gjersvik P. Weight-for-length, early weight-gain velocity and atopic dermatitis in infancy and at two years of age: a cohort study. BMC Pediatr. 2017 Jun 7;17(1):141. doi: 10.1186/s12887-017-0889-6. PMID 28592289
- [Derived] Rolfsjord LB, Bakkeheim E, Berents TL, Alm J, Skjerven HO, Carlsen KH, Mowinckel P, Sjobeck AC, Carlsen KCL. Morning Salivary Cortisol in Young Children: Reference Values and the Effects of Age, Sex, and Acute Bronchiolitis. J Pediatr. 2017 May;184:193-198.e3. doi: 10.1016/j.jpeds.2017.01.064. Epub 2017 Mar 8. PMID 28284475
- [Derived] Skjerven HO, Megremis S, Papadopoulos NG, Mowinckel P, Carlsen KH, Lodrup Carlsen KC; ORAACLE Study Group. Virus Type and Genomic Load in Acute Bronchiolitis: Severity and Treatment Response With Inhaled Adrenaline. J Infect Dis. 2016 Mar 15;213(6):915-21. doi: 10.1093/infdis/jiv513. Epub 2015 Oct 27. PMID 26508124
- [Derived] Skjerven HO, Rolfsjord LB, Berents TL, Engen H, Dizdarevic E, Midgaard C, Kvenshagen B, Aas MH, Hunderi JOG, Stensby Bains KE, Mowinckel P, Carlsen KH, Lodrup Carlsen KC. Allergic diseases and the effect of inhaled epinephrine in children with acute bronchiolitis: follow-up from the randomised, controlled, double-blind, Bronchiolitis ALL trial. Lancet Respir Med. 2015 Sep;3(9):702-708. doi: 10.1016/S2213-2600(15)00319-7. Epub 2015 Aug 25. PMID 26321593
- [Derived] Skjerven HO, Hunderi JO, Brugmann-Pieper SK, Brun AC, Engen H, Eskedal L, Haavaldsen M, Kvenshagen B, Lunde J, Rolfsjord LB, Siva C, Vikin T, Mowinckel P, Carlsen KH, Lodrup Carlsen KC. Racemic adrenaline and inhalation strategies in acute bronchiolitis. N Engl J Med. 2013 Jun 13;368(24):2286-93. doi: 10.1056/NEJMoa1301839. PMID 23758233
- See also: Oslo University Hospital — http://www.ous.no/